CLINICAL TRIAL: NCT03523130
Title: Application of IV 99mTc-tilmanocept for Imaging of Macrophage-specific Inflammation
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2018P000146
Record Dates: First submitted 2018-04-17; First posted 2018-05-14 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: HIV
Keywords: Macrophage-specific inflammation; Arterial inflammation; Neuroinflammation; SPECT/CT; Tilmanocept
MeSH Terms: conditions — Arteritis; Neuroinflammatory Diseases | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV-infected
  Interventions: Diagnostic Test: Imaging
- non-HIV-infected
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — Macrophage-specific inflammation

SUMMARY:
The purpose of this study is to evaluate uptake of intravenously administered 99mTc-tilmanocept using single photon emission computed tomography (SPECT/CT) scanning in individuals with HIV and individuals without HIV.

DETAILED DESCRIPTION:
People living with HIV (PLWH) have an increased risk of cardiovascular disease (CVD) compared to individuals without HIV. Increased systemic immune activation and arterial inflammation are thought to contribute to this increased risk by affecting the highly inflammatory process of atherosclerotic plaque formation and progression. This study will evaluate whether intravenous administration of a macrophage-specific imaging agent, 99mTc-tilmanocept, followed by SPECT/CT scanning can permit quantification of aortic 99mTc-tilmanocept uptake, reflective of aortic macrophage-specific inflammation among participants with HIV. We will also compare aortic 99mTc-tilmanocept uptake in participants with HIV to participants without HIV. Immunology parameters such as markers of immune activation and traditional CVD parameters will be assessed in relation to imaging assessments.

ELIGIBILITY:
HIV-infected participants:

Inclusion Criteria:

* men and women, ages 18 to 80, with documented HIV infection
* current use of antiretroviral therapy (ART), with no changes to regimen within last 3 months

Exclusion Criteria:

* pregnancy or breastfeeding
* known active opportunistic infection requiring ongoing medical therapy (not including Hepatitis B/C)
* CD4 count < 50 cells/mm3
* history of myocardial infarction,acute coronary syndrome, or coronary artery stenting or surgery
* stable or unstable angina
* recent and/or current treatment with prescription, systemic steroids or anti-inflammatory/immune suppressant medical therapies
* current use of statin or use of statin for > 1 month within the last 6 months
* known allergy to dextrans and/or DTPA and/or radiometals
* eGFR < 60 ml/min/1.73 m2 calculated by CKD-EPI
* known severe allergy to iodinated contrast media
* contraindication to nitroglycerin
* significant radiation exposure (>2 CT angiograms) received within the past 12 months
* reported active illicit drug use
* concurrent enrollment in another research study judged by the study investigators to interfere with the current study

Non-HIV-infected participant:

Inclusion criteria:

-men and women, ages 18 to 80, without HIV infection

Exclusion Criteria:

* pregnancy or breastfeeding
* history of myocardial infarction, acute coronary syndrome, or coronary artery stenting or surgery
* stable or unstable angina
* recent and/or current treatment with prescription, systemic steroids or anti-inflammatory/immune suppressant medical therapies
* current use of statin or use of statin for > 1 month within the last 6 months
* known allergy to dextrans and/or DTPA and/or radiometals
* eGFR < 60 ml/min/1.73 m2 calculated by CKD-EPI
* known severe allergy to iodinated contrast media
* contraindication to nitroglycerin
* significant radiation exposure (>2 CT angiograms) received within the past 12 months
* reported active illicit drug use
* concurrent enrollment in another research study judged by the study investigators to interfere with the current study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected participants and non-HIV-infected participants
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Aortic uptake of intravenously administered 99mTc tilmanocept on SPECT/CT | within 6 weeks of screening visit

SECONDARY OUTCOMES:
Aortic plaque burden and morphology on CT angiography | within 6 weeks of screening visit
  Aortic plaque burden and morphology will be assessed through measurement of total, calcified, and non-calcified aortic plaque volume (mm3).
Traditional markers of cardiovascular disease (CVD) risk in relation to cardiovascular imaging outcomes | within 6 weeks of screening visit
  We will calculate a risk score of future CVD risk (%) which will take into account traditional markers of CVD risk such as blood pressure, lipid levels, and age.
Inflammatory markers in relation to cardiovascular imaging outcomes | within 6 weeks of screening visit
  The following inflammatory markers will be evaluated: soluble CD163 (ng/ml) , soluble CD 14 (ng/ml) , and Lp-PLA2 (ng/ml).
Imaging assessments of the coronary vasculature | within 6 weeks of screening visit
  Cardiac CT angiography will be used to assess the coronary vasculature. Total, calcified, and non-calcified coronary plaque volume (mm3) will be measured.
Comparison of imaging assessments between HIV-infected participants and non-HIV-infected participants | within 6 weeks of screening visit
  We will compare the standardized uptake values on SPECT/CT of HIV-infected participants and non-HIV-infected participants.
Uptake of intravenously administered 99mTc tilmanocept on SPECT/CT in regions other than the aorta | within 6 weeks of screening visit
  Uptake of tilmanocept on SPECT/CT will determined by calculating a standardized uptake value.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States